CLINICAL TRIAL: NCT02968602
Title: Minocycline and Tobacco Craving in Smokers With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deanna Kelly, Professor, Chief Treatment Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HP-00072110; 4K23DA034034-04 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia; Tobacco Use
MeSH Terms: conditions — Schizophrenia; Tobacco Use | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocycline (Experimental): Participants will take 50 mg minocycline capsules twice daily for 1 week, then take 100 mg capsules twice daily for 1 week.
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Participants will take capsules that match active drug, but contain no active ingredients, twice daily for week 1, and then will take capsules that match active drug, but contain no active ingredients, twice daily for week 2.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Minocycline — Minocycline capsules taken twice daily for two weeks.
  Arms: Minocycline
Other: Placebo — Placebo capsules taken twice daily for two weeks.
  Arms: Placebo

SUMMARY:
Craving for cigarettes is an important aspect that leads to challenges with smoking cessation. Persons with schizophrenia are more likely to smoke and to be heavier smokers than persons without schizophrenia, and may experience craving differently as well. Minocycline is an antibiotic medication that may impact craving. We will conduct a two-week randomized, double-blind, placebo-controlled, parallel group pilot study to investigate the effects of minocycline vs. placebo on craving and smoking behaviors in smokers with schizophrenia. Participants will take minocycline or matching placebo for two weeks. Participants will be assessed on aspects of craving and smoking behavior at baseline and after 1 and 2 weeks of minocycline or placebo treatment.

DETAILED DESCRIPTION:
Nicotine dependence is high in schizophrenia; nearly three times more prevalent than the general population. In smokers with schizophrenia, the risk of all-cause mortality is doubled and cardiovascular mortality risk is twelvefold higher than nonsmokers. Many factors influence smoking in persons with schizophrenia, but predictors of craving and smoking behavior are not well established. Craving is a major contributor to smoking behaviors, and, importantly, is a predictor of relapse risk. Since craving may precede relapse, it can be advantageous as a screening tool for those attempting cessation. In addition, focusing on treatments aimed to reduce craving may lead to better therapeutic targets. Minocycline may affect craving, perhaps due to inhibition of nitric oxide (NO) formation, as NO acts as a second messenger for glutamate and dopamine receptors. NO also facilitates the effects of nicotine in the reward circuit, and blockade of NO has been demonstrated to eliminate nicotine abstinence symptoms in rats. A small study has demonstrated that minocycline reduces cigarette craving in human subjects without severe mental illness. The investigators will conduct a two-week randomized, double-blind, placebo-controlled, parallel group pilot study to investigate the effects of minocycline vs. placebo on craving and indicators of smoking intensity in smokers with schizophrenia. Participants will take minocycline up to 200 mg daily or matching placebo for two weeks. Participants will complete cigarette cue-elicited craving platforms and related assessments at baseline, and after 1 and 2 weeks of minocycline or placebo treatment.

ELIGIBILITY:
Inclusion Criteria

* DSM-IV or DSM-5 diagnosis of schizophrenia or schizoaffective disorder
* Male or Female
* Age: 18 to 65 years
* Caucasian or Non-Caucasian
* Smoke at least 10 cigarettes daily
* Urine cotinine level ≥ 100 ng/ml (NicAlert® reading ≥ 3)
* Agrees to wear a head mounted display (HMD) for up to 45 minutes
* Able to complete the Evaluation to Sign Consent (ESC) with minimum score of 80%

Exclusion Criteria

* History of organic brain disease
* DSM-IV diagnosis of Alcohol or Substance Dependence within the last six months (except nicotine) or DSM-5 diagnosis of Substance Use Disorder in the last six months (except nicotine)
* DSM-IV diagnosis of Alcohol or Substance Abuse within the last one month (except nicotine) or DSM-5 diagnosis of Substance Use Disorder in the last six months (except nicotine)
* Pregnancy or lactation
* Severe liver dysfunction (LFT 3X upper limit of normal)
* Previous known hypersensitivity to tetracyclines
* Current treatment with tetracycline or derivative
* Treatment with oral contraceptives (unless a second form of birth control is used and documented)
* Treatment with cholestyramine or colestipol
* Treatment with Urinary alkalinizers (e.g., sodium lactate, potassium citrate)
* Treatment with warfarin
* Treatment with bupropion, varenicline, or nicotine replacement products in the month prior to study inclusion
* Less than two months treatment of adjunctive medications AND less than one month on same dose: beta blockers, antidepressants, mood stabilizers, antianxiety medications.
* Medical condition whose pathology or treatment would significantly increase the risk associated with the proposed protocol.
* History of head injury, seizures, or stroke
* Positive urine toxicology screen for substances of non-therapeutic use prior to craving assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psyciatric Research Center, Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This study was funded prior to the NIH requirements for sharing of IPD, therefore is not within our budget.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.43 (11.32) | 43.38 (8.22) | 43.4 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 6 | 5 | 11
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire for Smoking Urges-Brief
Description: This is a 10-item assessment used to measure craving to smoke and used in studies of smokers with schizophrenia. This scale has a score range from 0-100The change in QSU-Brief craving scores between time points (baseline to week 1, and baseline to week 2) will be assessed. The change in scores between the two timepoints will be calculated. The higher the score the stronger the urge to smoke is.
Time Frame: Baseline, Week 1, and Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline to week 1 | 42.1429 (16.23319) | 38.6429 (18.46663)
  Baseline to week 2 (Endpoint) | 43.4286 (18.03720) | 36.8571 (17.81467)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 7/16 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=16) | Placebo (N=16)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Arthritus (General disorders) | 1 (1) | 0 (0)
Hypersalavation (General disorders) | 0 (0) | 2 (5)
Sedation (General disorders) | 2 (2) | 3 (3)
Restlessness (General disorders) | 2 (3) | 0 (0)
Loss of Appetite (General disorders) | 2 (2) | 0 (0)
Insomnia (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stiffness (General disorders) | 1 (1) | 0 (0)
Uticaria (General disorders) | 1 (1) | 0 (0)
Somatic Concern (General disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Hostility (General disorders) | 1 (1) | 0 (0)
Tremor (General disorders) | 1 (1) | 0 (0)
"Zoning out" (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02968602/Prot_SAP_000.pdf